CLINICAL TRIAL: NCT01459367
Title: A Phase 3, Randomized, Double-Blind, Multicenter Study to Evaluate the Efficacy and Safety of TAK-438 (10 mg or 20 mg Once-Daily) Compared to AG-1749 (15 mg Once-Daily) in a 24-week Maintenance Treatment in Patients With Healed Erosive Esophagitis (EE).
Brief Title: Efficacy of TAK-438 Compared to AG-1749 (Lansoprazole) in the Maintenance Treatment of Healed Erosive Esophagitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-438/CCT-003; U1111-1125-1054 (Registry Identifier: WHO); JapicCTI-111662 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2011-10-24; First posted 2011-10-25 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Erosive Esophagitis
Keywords: Drug Therapy
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TAK-438 10 mg QD (Experimental)
  Interventions: Drug: TAK-438
- TAK-438 20 mg QD (Experimental)
  Interventions: Drug: TAK-438
- Lansoprazole 15 mg QD (Active Comparator)
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: TAK-438 — In the treatment period, the participants will receive treatment of TAK-438 20 mg, tablets, orally, once daily for up to 8 weeks.
  In the maintenance treatment period, the participants will receive treatment of TAK-438 10 mg, tablets, orally, once daily and lansoprazole placebo-matching capsules, orally, once daily for up to 24 weeks.
  Arms: TAK-438 10 mg QD
Drug: TAK-438 — In the treatment period, the participants will receive treatment of TAK-438 20 mg, tablets, orally, once daily for up to 8 weeks.
  In the maintenance treatment period, the participants will receive treatment of TAK-438 20 mg, tablets, orally, once daily and lansoprazole placebo-matching capsules, orally, once daily for up to 24 weeks.
  Arms: TAK-438 20 mg QD
Drug: Lansoprazole — In the treatment period, the participants will receive treatment of TAK-438 20 mg, tablets, orally, once daily for up to 8 weeks.
  In the maintenance treatment period, the participants will receive treatment of TAK-438 placebo-matching tablets, orally, once daily and lansoprazole 15 mg, capsules, orally, once daily for up to 24 weeks.
  Other Names: AG-1749
  Arms: Lansoprazole 15 mg QD

SUMMARY:
The purpose of this study is to confirm the efficacy of TAK-438, once daily (QD), compared to lansoprazole for the maintenance treatment of healed erosive esophagitis and to determine the clinical dose.

ELIGIBILITY:
Inclusion Criteria:

1. At Visit H-1 (start of the treatment period), the participants must have endoscopically confirmed erosive esophagitis of Grade A to D, as defined by the LA classification grading system, and the target number of participants who are clearly Grade C or D is 15% or more of the total participants.
2. Outpatients (including inpatient for examination)
3. Participants must have successfully completed the treatment period and have endoscopically healed EE at Week 2, 4, or 8 in the treatment period. Endoscopically healed EE is defined as those participants who have endoscopically confirmed EE of Grade O as defined by the LA classification grading system.

Exclusion Criteria:

1. Participants with an esophagus-related complication (eosinophilic esophagitis, esophageal varices, scleroderma, viral or fungal infection, esophageal stenosis, etc.), a history of radiotherapy or cryotherapy of the esophagus, a caustic or physiochemical trauma (esophageal sclerotherapy, etc.). However, participants with Schatzki's ring (mucosal tissue ring around inferior esophageal sphincter) or Barrett's esophagus are allowed to be included.
2. Participants who have received surgery or treatment affecting gastroesophageal reflux (cardioplasty, dilation of esophageal stenosis [excluding Schatzki's ring], etc.), or who have a history of surgery of stomach or duodenum (excluding removal of benign polyp under endoscopy)
3. Participants who have acute upper gastrointestinal bleeding, gastric or duodenal ulcer (mucosal defect with white coating) within 30 days prior to Visit H-1 (initiation of study drug administration). However, participants with gastric or duodenal erosions are allowed to be included.
4. Participants with a previous or current history of Zollinger-Ellison syndrome, or other gastric acid hypersecretion disorder

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2011-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Endoscopically confirmed recurrence rate of erosive esophagitis after 24 weeks of maintenance treatment | 24 Weeks.
  Endoscopic recurrence of erosive esophagitis is defined as those participants who have endoscopically confirmed EE of Grade A to D as defined by the Los Angeles (LA) Classification Grading System. The definitions of each grade are: Grade O (No mucosal break), Grade A (Mucosal break <5 mm), Grade B (Mucosal break ≥5 mm), Grade C (Mucosal break continuous between two or more folds and <75% of the circumference) and Grade D (Mucosal break ≥75% of the circumference).

SECONDARY OUTCOMES:
Endoscopically confirmed recurrence rate of erosive esophagitis after 12 weeks of maintenance treatment | 12 Weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Senior Manager, Study Director — Takeda
Locations (37):
- Japan (37):
  - Kashiwa-shi, Chiba
  - Yachiyo-shi, Chiba
  - Saijo-shi, Ehime
  - Fukuoka, Fukuoka
  - Kasuya-gun, Fukuoka
  - Koriyama-shi, Fukushima
  - Takayama-shi, Gifu
  - Annaka-shi, Gunma
  - Asahikawa-shi, Hokkaido
  - Sapporo, Hokkaido
  - Itami-shi, Hyōgo
  - Kobe, Hyōgo
  - Nishinomiya-shi, Hyōgo
  - Fujisawa-shi, Kanagawa
  - Yokohama, Kanagawa
  - Kochi, Kochi
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Sendai, Miyagi
  - Nagasaki, Nagasaki
  - Kishiwada-shi, Osaka
  - Osaka, Osaka
  - Suita-shi, Osaka
  - Takatsuki-shi, Osaka
  - Saga, Saga-ken
  - Kumagaya-shi, Saitama
  - Saitama-shi, Saitama
  - Tokorozawa-shi, Saitama
  - Bunkyo-ku, Tokyo
  - Chuo-ku, Tokyo
  - Hachioji-shi, Tokyo
  - Kokubunji-shi, Tokyo
  - Shibuya-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Toshima-ku, Tokyo
  - Shimonoseki-shi, Yamaguchi
  - Tsuru-shi, Yamanashi